CLINICAL TRIAL: NCT05341843
Title: Effectiveness of Sertraline in Alleviating Uremic Pruritis in Hemodialysis Patients
Brief Title: Sertraline Effect in Uremic Pruritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sertraline and uremic pruritis
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Uremic Pruritis
Keywords: sertraline, hemodialysis
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: This research is a double-blinded randomized multicentric clinical trial in which 50 haemodialysis patients will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
  * Group A: 25 patients will receive sertraline at the intended dose of 50 mg twice daily for 8 weeks.
  * Group B: 25 patients will receive a placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: a double blinded study as participants, health care providers as well as the outcome assessor will be unaware about the type of treatment each patient receive.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sertraline (Experimental): they will receive sertraline at the intended dose of 50 mg twice daily for 8 weeks.
  Interventions: Drug: sertraline
- placebo (Placebo Comparator): They will receive a placebo in the form of multivitamin tablets similar to the experimental drug with the same regimen, as one tablet /day for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: sertraline — sertraline at the intended dose of 50 mg twice daily for 8 weeks.
  Arms: sertraline
Drug: placebo — a placebo in the form of multivitamin tablets similar to the experimental drugs with the same regimen (one tablet /day for 8 weeks)
  Arms: placebo

SUMMARY:
This study aims to assess the effect of sertraline on uremic pruritis in patients undergoing regular haemodialysis.

DETAILED DESCRIPTION:
The reported prevalence of uremic pruritus in adult hemodialysis patients has varied over the years, and some studies suggest the prevalence may be decreasing with more effective dialysis. One of the largest trials (the Dialysis Outcomes and Practice Patterns Study [DOPPS]) reported that the prevalence of moderate pruritus remained constant at 18 percent until 2015.

A direct role for proinflammatory T cells and cytokines is suggested by studies that showed higher levels of proinflammatory T helper-1 (TH1) cells, C-reactive protein, interleukin-6, and interleukin-2 levels among hemodialysis patients versus those without pruritus. Also, histamine release from mast cells, other pruritogens and xerosis have been all implicated in the pathogenesis of uremic pruritus.

Less convincing associations have also been made to anemia, male sex, increased beta-2 microglobulin levels, serotype human leukocyte antigen (HLA)-B35, and comorbidities including congestive heart failure and neurologic disease. The risk of uremic pruritis appears to be independent of ethnicity, type of dialysis, and underlying renal disease. No single cause underlying uremic pruritus has been identified. Multiple factors have been associated in observational studies, and supportive therapies that are used to treat uremic pruritus have targeted such factors.

High quality evidence on which to base recommendations for the treatment of uremic pruritus is limited. Many pharmacologic treatments have been proposed for uremic pruritis through different clinical trials. However, the results were quite variable and most of these studies were small uncontrolled trials and hence they were flawed.

Several studies have revealed that the selective serotonin reuptake inhibitors (SSRI) could reduce the severity of pruritus. Sertraline hydrochloride is a selective serotonin reuptake inhibitor which established improvement in itching in patients with cholestatic pruritis. This was supported by Browning et al. (2003) whose study showed 86% of subjects who had been given sertraline for another indication improved considerably with pruritus disappearing in 30% of the subjects.

Generally, most of the previous research has tended to focus on cholestatic pruritis rather than uremic pruritis. Although enough is known to determine a reasonable approach to a patient with uremic pruritus, more research is needed to understand the pathophysiology of this condition and to establish more reliable treatments. Hence, this study is organized in an attempt to find out the effect of sertraline on alleviation of uremic pruritus.

ELIGIBILITY:
Inclusion Criteria:

1. ≥1 month of maintenance haemodialysis, 3 times per week for 4 hours.
2. Adult patients with ages between 18-80 years.

Exclusion Criteria:

1. Primary skin diseases (eczema, psoriasis, allergic dermatitis or drug rash).
2. Peripheral neuropathy, thyroid disease, leukemia, lymphoma, liver disease, Systemic lupus erythematosus or pregnancy.
3. Patients who consumed emollients cream, antihistamine, opioid antagonist, immunosuppressants, cholestyramine, corticosteroids or UVB phototherapy 1 month before study.
4. calcium X phosphorus (Ca X P) >55.0 mg/dl, P >5.5 mg/dl, parathyroid hormone (PTH) >450 pg/ml.
5. Selective serotonin reuptake inhibitors intolerance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
change in uremic pruritis intensity | 8 weeks
  Assessment of pruritis will be done before and after the course of treatment (8 weeks) through the following scores:
  I) Visual analogue scale (VAS) II) 5D itch scale

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; Sherif aziz Zaki, MD, Study Chair — professor; Iman ezzat El Gohary, MD, Study Chair — professor; Heidi Hesham Abd El Hamid, MBBCh, Study Chair — Resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patel TS, Freedman BI, Yosipovitch G. An update on pruritus associated with CKD. Am J Kidney Dis. 2007 Jul;50(1):11-20. doi: 10.1053/j.ajkd.2007.03.010. PMID 17591521
- [Background] Pisoni RL, Wikstrom B, Elder SJ, Akizawa T, Asano Y, Keen ML, Saran R, Mendelssohn DC, Young EW, Port FK. Pruritus in haemodialysis patients: International results from the Dialysis Outcomes and Practice Patterns Study (DOPPS). Nephrol Dial Transplant. 2006 Dec;21(12):3495-505. doi: 10.1093/ndt/gfl461. Epub 2006 Sep 12. PMID 16968725
- [Background] Pauli-Magnus C, Mikus G, Alscher DM, Kirschner T, Nagel W, Gugeler N, Risler T, Berger ED, Kuhlmann U, Mettang T. Naltrexone does not relieve uremic pruritus: results of a randomized, double-blind, placebo-controlled crossover study. J Am Soc Nephrol. 2000 Mar;11(3):514-519. doi: 10.1681/ASN.V113514. PMID 10703675
- [Background] Rayner HC, Larkina M, Wang M, Graham-Brown M, van der Veer SN, Ecder T, Hasegawa T, Kleophas W, Bieber BA, Tentori F, Robinson BM, Pisoni RL. International Comparisons of Prevalence, Awareness, and Treatment of Pruritus in People on Hemodialysis. Clin J Am Soc Nephrol. 2017 Dec 7;12(12):2000-2007. doi: 10.2215/CJN.03280317. Epub 2017 Sep 18. PMID 28923831
- [Background] Kimmel M, Alscher DM, Dunst R, Braun N, Machleidt C, Kiefer T, Stulten C, van der Kuip H, Pauli-Magnus C, Raub U, Kuhlmann U, Mettang T. The role of micro-inflammation in the pathogenesis of uraemic pruritus in haemodialysis patients. Nephrol Dial Transplant. 2006 Mar;21(3):749-55. doi: 10.1093/ndt/gfi204. Epub 2005 Oct 25. PMID 16249205
- [Background] Fallahzadeh MK, Roozbeh J, Geramizadeh B, Namazi MR. Interleukin-2 serum levels are elevated in patients with uremic pruritus: a novel finding with practical implications. Nephrol Dial Transplant. 2011 Oct;26(10):3338-44. doi: 10.1093/ndt/gfr053. Epub 2011 Mar 3. PMID 21372257
- [Background] Charlesworth EN, Beltrani VS. Pruritic dermatoses: overview of etiology and therapy. Am J Med. 2002 Dec 16;113 Suppl 9A:25S-33S. doi: 10.1016/s0002-9343(02)01434-1. PMID 12517579
- [Background] Stander S, Bockenholt B, Schurmeyer-Horst F, Weishaupt C, Heuft G, Luger TA, Schneider G. Treatment of chronic pruritus with the selective serotonin re-uptake inhibitors paroxetine and fluvoxamine: results of an open-labelled, two-arm proof-of-concept study. Acta Derm Venereol. 2009;89(1):45-51. doi: 10.2340/00015555-0553. PMID 19197541
- [Background] Mayo MJ, Handem I, Saldana S, Jacobe H, Getachew Y, Rush AJ. Sertraline as a first-line treatment for cholestatic pruritus. Hepatology. 2007 Mar;45(3):666-74. doi: 10.1002/hep.21553. PMID 17326161
- [Background] Snit M, Gawlik R, Lacka-Gazdzik B, Kuzniewicz R, Dwornicki M, Owczarek A, Walaszczyk M, Grabiec P, Grzeszczak W. Substance P and intensity of pruritus in hemodialysis and peritoneal dialysis patients. Med Sci Monit. 2013 Sep 2;19:723-32. doi: 10.12659/MSM.889349. PMID 23995243
- [Background] Ko MJ, Wu HY, Chen HY, Chiu YL, Hsu SP, Pai MF, Ju-Yehyang, Lai CF, Lu HM, Huang SC, Yang SY, Wen SY, Chiu HC, Hu FC, Peng YS, Jee SH. Uremic pruritus, dialysis adequacy, and metabolic profiles in hemodialysis patients: a prospective 5-year cohort study. PLoS One. 2013 Aug 6;8(8):e71404. doi: 10.1371/journal.pone.0071404. Print 2013. PMID 23940749
- [Background] Wu HY, Peng YS, Chen HY, Tsai WC, Yang JY, Hsu SP, Pai MF, Lu HM, Chiang JF, Ko MJ, Wen SY, Chiu HC. A Comparison of Uremic Pruritus in Patients Receiving Peritoneal Dialysis and Hemodialysis. Medicine (Baltimore). 2016 Mar;95(9):e2935. doi: 10.1097/MD.0000000000002935. PMID 26945400
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Derived] Elsayed MM, Elgohary IE, Abdelhamid HHS, Zaki SA. The effectiveness of sertraline in alleviating uremic pruritus in hemodialysis patients: a randomized clinical trial. BMC Nephrol. 2023 Jun 3;24(1):155. doi: 10.1186/s12882-023-03212-3. PMID 37270517